CLINICAL TRIAL: NCT04739878
Title: Prospective Study On Novel Usage of Airway Ultrasound To Detect Subglottic Secretion Above Endotracheal Tube(ETT) Cuff
Brief Title: SUBSUS (SUBglottic Secretion at Ultrasound Score)
Acronym: SUBSUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Raja Permaisuri Bainun (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 58284
Record Dates: First submitted 2021-01-18; First posted 2021-02-05 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Ventilator Associated Pneumonia
Keywords: subglottic secretion; airway ultrasound; ventilator associated pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound Airway (Experimental): Ultrasound Airway for subglottic secretion
  Interventions: Procedure: Airway Ultrasound

INTERVENTIONS:
Procedure: Airway Ultrasound — Comparison between Airway ultrasound and CT cervical
  Other Names: Cervical CT plain

SUMMARY:
To compare the performance of ultrasound in detecting subglottic secretion above the ETT tube cuff in comparison to computed tomography (CT) scan.

DETAILED DESCRIPTION:
Airway ultrasound will be performed at the bedside prior to CT scan in all intubated patients who fulfiled the criteria. The image of subglottic secretion was then compared to the plain CT cervical. The findings of the CT was examined by a radiologist.

ELIGIBILITY:
Inclusion Criteria:

* age more than 18 years old
* ETT in situ
* indicated for CT cervical scan

Exclusion Criteria:

* neck subcutaneous emphysema
* neck scar or surgical dressing around the neck which can lead to difficulty in obtaining an optimal ultrasound image.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Prospective Study on Novel Usage of Airway Ultrasound To Detect Subglottic Secretion Above Endotracheal Tube Cuff | 90 days
  Compare the performance of airway ultrasound and cervical CT scan to diagnose subglottic secretion.

CONTACTS AND LOCATIONS:
Overall Officials: Adi Osman, MD, Principal Investigator — Hospital Raja Permaisuri Bainun
Locations (1):
- Raja Permaisuri Bainun Hospital, Ipoh, Perak, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adi O, Fong CP, Sallehuddin RM, Ahmad AH, Sum KM, Yusof ZM, Via G, Tavazzi G. Airway ultrasound to detect subglottic secretion above endotracheal tube cuff. Ultrasound J. 2023 May 6;15(1):23. doi: 10.1186/s13089-023-00318-5. PMID 37148375

DOCUMENTS (1):
  • Study Protocol (2021-01-31): https://cdn.clinicaltrials.gov/large-docs/78/NCT04739878/Prot_000.pdf